CLINICAL TRIAL: NCT04674007
Title: The Effect of Cognitive Dual Task and Mental Fatigue on Landing Biomechanics
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000525-2
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Landing Biomechanics; Fatigue
Keywords: landing; biomechanics; fatigue; dual task
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy basketball, volleyball and handball players: Healthy basketball, volleyball and handball players
  Interventions: Other: 3D analysis of landing task

INTERVENTIONS:
Other: 3D analysis of landing task — Landing tasks (anticipated, unanticipated and cognitive dual task) are investigated with 3D analysis by using an opto-electronic system

SUMMARY:
In this study, three-dimensional biomechanics , by means of lower limb joint angles and moments (opto-electronic system with synchronised force plate), of landing tasks (anticipated, unanticipated and cognitive dual task) before and after a mental fatigue protocol will be compared in a population of basketball, handball and volleyball players.

DETAILED DESCRIPTION:
In this study, three-dimensional biomechanics , by means of lower limb joint angles and moments (opto-electronic system with synchronised force plate), of landing tasks (anticipated, unanticipated and cognitive dual task) before and after a mental fatigue protocol will be compared in a population of basketball, handball and volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* volleyball, basketball of handball players
* male

Exclusion Criteria:

* history or surgery of the lower extremities
* history of fractures of the lower extremities

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volleyball, basketball and handball players
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Joint angles lower extremity | The same day/test moment, immediately after fatiguing exercises
  Joint angles will be extracted with an opto-electronic system and synchronised force plate
Joint moments lower extremity | The same day/test moment, immediately after fatiguing exercises
  Joint moments will be extracted with an opto-electronic system and synchronised force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Roel De Ridder, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided